CLINICAL TRIAL: NCT00791076
Title: The Effect of Pancreatic Polypeptide on Insulin Requirements for Type 1 (Auto-immune) and Post-pancreatectomy Diabetic Patients
Brief Title: The Effect of Pancreatic Polypeptide on Insulin Requirements for Type 1 & Post-pancreatectomy Diabetic Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left JHU
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00010957
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Insulin pump therapy; Type 1 diabetic; Chronic pancreatitis; Pancreatic resection; Pancreatic polypeptide
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Pancreatitis, Chronic | interventions — Sodium Chloride; Pancreatic Polypeptide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline Placebo (Placebo Comparator): Saline
  Interventions: Drug: Placebo
- Pancreatic Polypeptide (Active Comparator): Pancreatic Polypeptide
  Interventions: Drug: Pancreatic Polypeptide (PP)

INTERVENTIONS:
Drug: Placebo — 2pmol/kg-1/min-1 placebo infused continuously over 72 hours.
  Other Names: Saline
  Arms: Saline Placebo
Drug: Pancreatic Polypeptide (PP) — 2pmol/kg-1/min-1 PP infused continuously over 72 hours.
  Other Names: PP
  Arms: Pancreatic Polypeptide

SUMMARY:
The goal of this research is to see if pancreatic polypeptide (PP), a hormone that is naturally produced by the pancreas and that works to control the amount of glucose that the liver makes, will reduce the amount of insulin required for people who must take insulin to maintain their normal blood glucose level.

DETAILED DESCRIPTION:
The pancreas is a large gland located behind the stomach. One of the functions of the pancreas is to produce two hormones: insulin and pancreatic polypeptide. Insulin helps the cells to take in glucose. The liver makes glucose and insulin normally acts to decrease or shut off the liver's production of glucose. However, in patients whose pancreas no longer makes insulin or makes low levels of pancreatic polypeptide the liver cannot perform these duties as well. Studies have shown that these important functions of the liver are improved for these patients when pancreatic polypeptide is given together with their insulin. Because PP increases the liver's sensitivity to insulin and thereby reduces the amount of glucose produced by the liver, this will result in fewer swings in blood sugar levels both in the upper and lower range. With fewer swings in blood glucose, a patient should decrease the amount of insulin used. One of the main benefits of lowering total insulin requirement is a reduction in the development of dangerous low blood sugar levels.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers between the ages of 18-75 with:
* 10 subjects who are status post pancreatic resection and 10 volunteers who are Type 1 diabetic for > 8 years (volunteers must have a stable glycemic profile that includes use of an insulin pump to control their blood glucose) with or without prior pancreatic resection.
* HbA1c levels ≤ 8.5.

Exclusion Criteria:

* Lactating or pregnant females.
* Brittle or Labile diabetics: Volunteers with extremely erratic patterns of glucose control with large fluctuations in glucose levels for no obvious reason.
* Allergy to beef or beef by-products.
* Hypoglycemia within the past year requiring medical or other assistance to correct.
* Known autonomic neuropathy.
* Documented blood glucose under 60 mg within the past year and hypoglycemic unawareness.
* Durations of type 1 Diabetes Melitis (DM) ≤ 8 years.
* Not currently on pump therapy.
* Type 1 DM who has a BMI ≥ 35.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Elahi, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Saline
  Placebo: 2pmol/kg-1/min-1 PP or placebo infused continuously over 72 hours.
  OR
  Pancreatic Polypeptide
  Pancreatic Polypeptide (PP): 2pmol/kg-1/min-1 PP or placebo infused continuously over 72 hours.
Period: Overall Study
Arm/Group | All Participants
Started | 8
Completed | 0
Not Completed | 8
Not completed — Study was terminated,PI left institution | 8

BASELINE CHARACTERISTICS:
Population: This study was terminated prematurely when the PI left the institution. Although 8 participants were enrolled in this study, their assignment to Arm/Group is unknown, since no data are available.
Groups:
- All Study Participants: 2pmol/kg-1/min-1 saline infused continuously over 72 hours OR
  2pmol/kg-1/min-1 PP infused continuously over 72 hours.
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Customized [Number; unit: participants]
  >=18 and <=75 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Total Amount of Insulin Administered While on Placebo/PP.
Description: Glucose values and the pattern of glycemic excursions over the 72 hour test period.
Time Frame: 2 years
Population: Data was not collected for this outcome measure. The P.I. left the institution and the study was terminated.
Groups:
- Saline Placebo: Saline
  Placebo: 2pmol/kg-1/min-1 PP or placebo infused continuously over 72 hours.
- Pancreatic Polypeptide: Pancreatic Polypeptide
  Pancreatic Polypeptide (PP): 2pmol/kg-1/min-1 PP or placebo infused continuously over 72 hours.
Arm/Group | Saline Placebo | Pancreatic Polypeptide
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Frequency of Hypoglycemia Defined as < 60 mg/dl.
Time Frame: 72 hours
Population: The PI left the institution and this study was terminated due to noncompliance with our Institutional Review Board. Data, if collected,is unknown since no data are available.
Arm/Group | Saline Placebo | Pancreatic Polypeptide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The PI left the institution and this study was terminated due to noncompliance with our Institutional Review Board. Time frame for Adverse event data, if collected, is unknown since no data are available.
Description: The PI left the institution and this study was terminated due to noncompliance with our Institutional Review Board. Adverse event data, if collected, is unknown since no data are available.
Arm/Group | Saline Placebo | Pancreatic Polypeptide
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes